CLINICAL TRIAL: NCT02063334
Title: The Effect of a High-dose Oral Vitamin D3 Bolus on Serum 25-hydroxyvitamin D3 and Vitamin D Receptor Target Gene Expression (VitDbol)
Brief Title: The Effect of a High-dose Oral Vitamin D3 Bolus on Serum 25(OH)D3 and Vitamin D Receptor Target Gene Expression
Acronym: VitDbol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VitDbol
Record Dates: First submitted 2014-02-04; First posted 2014-02-14 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-06

CONDITIONS: Vitamin D Receptor Target Gene Expression; Serum 25(OH)D Concentration
Keywords: vitamin D3; cholecalciferol; calcidiol; 25-hydroxyvitamin D; gene expression; vitamin D receptor; randomized controlled trial; men; adults
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 (Active Comparator): 2000 micrograms of vitamin D3 in two doses during one day
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Placebo in two doses during one day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — In total 25 pills will be taken by the subjects, each containing 80 micrograms of vitamin D3 or placebo. Of the 25 pills, 13 will be taken in the morning with breakfast and 12 with lunch.
  Other Names: cholecalciferol
  Arms: Vitamin D3
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate whether a high-dose vitamin D3 oral bolus (2000 micrograms) produces marked vitamin D receptor target gene expression response and whether there is large inter-individual variation.

DETAILED DESCRIPTION:
Serum 25-hydroxyvitamin D [25(OH)D3] is a well-established marker for vitamin D status of the human body. In addition to the general importance of vitamin D for bone health, low serum 25(OH)D3 concentrations have been associated with increased risk of several health outcomes, such as autoimmune diseases, type 2 diabetes and cardiovascular complications. However, there is significant inter-individual variation in the average serum 25(OH)D3 concentrations and also in the response to supplementation with vitamin D. Genetic and epigenetic factors have been suggested to be responsible for a large part of the variation, but currently there is little information about the health effects of the variation.

In our previous study (VitDmet, Clinicaltrials.gov NCT01479933) we showed that only half of the participants responded to the 5-month vitamin D3 supplementation of 40 µg/day or 80 µg/day as expected and that certain vitamin D receptor (VDR) target genes were suitable biomarkers for displaying the transcriptomic response of human tissues to vitamin D3 supplementation.

The purpose of the current study is to investigate whether a high-dose vitamin D3 oral bolus produces marked VDR target gene expression response and whether there is large inter-individual variation, as what was suggested with the 5-month lower-dose supplementation.

In the Trial 1, the subjects are randomized to receive either 2,000 micrograms (80 000 IU) of vitamin D3 (n=20) or placebo (n=10) in one day. Blood samples are collected for peripheral blood mononuclear cell isolation and serum 25(OH)D3 measurements at baseline and 24 h and 48 h and 30 days after the first dose. Blood samples are also collected for immunomarker analyses. In the Trial 2, the procedures of the Trial 1 are repeated in two subjects with known low and high serum 25(OH)D3 concentrations in order to investigate more specifically the impact of different starting levels of serum 25(OH)D3.

In February 2015, new subjects were recruited to enter the Trial 1 in order to increase the size of the study. All the new subjects received the 2,000 microgram bolus of vitamin D3, there were no new subjects in the placebo arm.

June 30, 2016. Change to protocol: There will be no Trial 2, but instead the blood samples obtained in the Trial 1 from up to six subjects will be used for the additional analyses. The subjects are selected based on the response to vitamin D supplementation in the Trial 1.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking
* BMI 20-25 kg/m2.

Exclusion Criteria:

* History of kidney stones, renal failure or dialysis, hypercalcemia, hypo- or hyperparathyroidism, severe liver disease (cirrhosis), or sarcoidosis or other granulomatous diseases, such as active chronic tuberculosis or Wegener's granulomatosis.
* Continuous use of anti-inflammatory medicines.
* Regular use of supplements containing vitamin D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vitamin D target gene expression | 24 h, 48 h, and 30 days after the baseline
  Effect of 2000 microgram vitamin D3 dose or placebo on the expression of vitamin D receptor target genes

SECONDARY OUTCOMES:
Change from baseline in serum 25(OH)D | 24 h, 48 h, and 30 days after the baseline
  Effect of 2000 microgram vitamin D3 dose or placebo on serum 25(OH)D3 concentrations

OTHER OUTCOMES:
Change from baseline in immunomarkers | 24 h, 48 h, and 30 days after the baseline
  Effect of 2000 microgram Vitamin D3 dose or placebo on immune system and inflammatory responses, such as hs-CRP, IL-6, TNF-alfa and IL-1RA.
Change from baseline in glucose metabolism | 24 h, 48 h, and 30 days after the baseline
  Effect of 2000 microgram vitamin D3 dose or placebo on glucose metabolism responses, i.e. blood glucose and insulin
Change from baseline in safety measurements | 48 h and 30 days after the baseline
  Serum calcium, alanine transaminase (ALAT), gamma-glutamyl transferase (GGT) and creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Jyrki K Virtanen, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

REFERENCES:
- [Derived] Seuter S, Virtanen JK, Nurmi T, Pihlajamaki J, Mursu J, Voutilainen S, Tuomainen TP, Neme A, Carlberg C. Molecular evaluation of vitamin D responsiveness of healthy young adults. J Steroid Biochem Mol Biol. 2017 Nov;174:314-321. doi: 10.1016/j.jsbmb.2016.06.003. Epub 2016 Jun 6. PMID 27282116